CLINICAL TRIAL: NCT04991051
Title: HRDx-Ovarian. A Cross-sectional, Noninterventional, Multicentre Study to Determine the Prevalence of Homologous Recombination Deficiency Among Women With Newly Diagnosed, High-grade, Serous or Endometrioid Ovarian, Primary Peritoneal, and/or Fallopian Tube Cancer.
Brief Title: Study to Determine the Prevalence of Homologous Recombination Deficiency Among Women With Newly Diagnosed, High-grade, Serous or Endometrioid Ovarian, Primary Peritoneal, and/or Fallopian Tube Cancer
Acronym: HALO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0818R00007
Record Dates: First submitted 2021-07-08; First posted 2021-08-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Fallopian Tube Cancer
Keywords: Cancer, HRD-testing, ovarian
MeSH Terms: conditions — Fallopian Tube Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
To maximise the accessibility and benefit of PARP inhibitors to eligible patients, it is essential to know the prevalence of HRD in women with advanced high-grade serous or endometrioid ovarian cancer. Presently, the prevalence data for HRD are available from selected geographies only and range from 31% to 50%. Furthermore, the risk factors associated with HRD and clinical characteristics of patients with HRD need exploration for region-specific differences. In the present study, we will estimate the region- and country-specific prevalence of HRD in women with stage III or IV high-grade serous or endometrioid ovarian, primary peritoneal, and/or fallopian tube cancer and associated risk factors with clinical characteristics in Asia-Pacific countries, Latin America, Africa, Russia, Australia, and Middle East countries.

The findings of the study will help the oncologists in optimal patient selection and clinical decision-making for the first-line maintenance of patients with HGSOC

DETAILED DESCRIPTION:
This cross-sectional, noninterventional, multicentre, epidemiological, observational study is designed to determine the prevalence of HRD in patients with newly diagnosed high-grade serous or endometrioid ovarian, primary peritoneal, and/or fallopian tube cancer. The study will also determine the prevalence of tBRCA1m/tBRCA2m, genomic instability, and identify the associated risk factors in several countries across broad geographic regions. The patients with newly diagnosed high-grade (stage III or IV of Federation of Gynecology and Obstetrics [FIGO] classification 2014, Prat J, 2015) ovarian cancer, having the availability of formalin-fixed paraffin-embedded (FFPE) archival tumour tissue block(s) collected within past 120 days will be screened to enrol a minimum of 405 women after obtaining written informed consent and eligibility assessment. The FFPE tumour tissue block(s) collected as part of routine clinical care at public or private ovarian cancer management and or diagnostic facilities in the selected countries will be sent for testing at Myriad Genetics laboratories Inc.

at Salt Lake City, United States of America (USA) through Myriad's local logistics network.

This study will have a single visit.

The study centres and the respective investigators will be selected through a site-level feasibility process after assessing the following:

* availability of the average number patients with newly diagnosed stage III and IV serous or endometrioid ovarian, primary peritoneal, and/or fallopian tube cancer.
* completeness of patient medical records pertaining to diagnostics and having the facility, capacity, and competence of collecting and archiving FFPE tumour tissue block(s).

Assessment and selection of study centres by the study sponsor AstraZeneca (AZ) will be an ongoing process during the entire course of the study until completion of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age or adults according to age of majority as defined by the local regulations;
* Willing and able to provide written informed consent for participation in the study;
* Patients with histologically confirmed new diagnosis (within past 120 days of enrolment) of high-grade (stage III or IV of FIGO classification 2014) serous or endometrioid ovarian, primary peritoneal, and/or fallopian tube cancer;
* Patients having availability of histopathology report and FFPE archival tumour tissue block(s) collected within past 120 days of enrolment.

Exclusion Criteria:

* Patients with mucinous, clear-cell, undifferentiated carcinoma or malignant Brenner's tumour;
* Patients diagnosed with any severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of the study results, and those in the judgment of the investigator are not appropriate for enrolment in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with high-grade (stage III or IV of FIGO classification 2014) ovarian cancer will be eligible for inclusion into the study if they meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
The overall percentage of patients diagnosed with positive HRD status | Baseline
  At baseline of this study

SECONDARY OUTCOMES:
Region- and country-specific percentages of patients with positive HRD status | Baseline
  At baseline of this study
Overall, region- and country-specific percentages of patients with tBRCA1m/tBRCA2m within each geographical region | Baseline
  At baseline of this study
Overall, region- and country-specific percentages of patients with GIS-positive status within each geographical region | Baseline
  At baseline of this study
Association of HRD-positive status and tBRCA1m/tBRCA2m | Baseline
  At baseline of this study

CONTACTS AND LOCATIONS:
Locations (24):
- Research Site, Kuwait City, Kuwait
- Research Site, Muscat, Oman
- Research Site, Doha, Qatar
- Russia (18):
  - Research Site, Balashikha, Moscow Oblast
  - Research Site, Istra Settlement, Moscow Oblast
  - Research Site, Kolomna, Moscow Oblast
  - Research Site, Arkhangelsk
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Tula
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Yaroslavl
  - Research Site, Yuzhno-Sakhalinsk
- Saudi Arabia (2):
  - Research Site, Jeddah
  - Research Site, Mecca
- Research Site, Alain, United Arab Emirates

REFERENCES:
- [Derived] Liou WS, Chao A, Sheu BC, Yeh LS, Wu CH. Prevalence of homologous recombination deficiency in ovarian, primary peritoneal, and/or fallopian tube cancer: results from HALO-Taiwan subset. J Gynecol Oncol. 2025 Dec 29. doi: 10.3802/jgo.2026.37.e55. Online ahead of print. PMID 41575336
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0818R00007&attachmentIdentifier=c5406519-b22f-4424-9a59-8e048f4f7f0b&fileName=CSR__D0818R00007_HALO_Final.v1.0_-_signed_Redacted.pdf&versionIdentifier=